CLINICAL TRIAL: NCT06540326
Title: Clinical Study of Second-line Treatment of Patients With Advanced Colorectal Cancer With Irinotecan Liposome (II), Fluorouracil in Combination With Bevacizumab or Cetuximab
Brief Title: Clinical Study of Second-line Treatment in Advanced Colorectal Cancer With Chemotherapy With Bevacizumab or Cetuximab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-CRC-II-012
Record Dates: First submitted 2024-07-22; First posted 2024-08-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — irinotecan sucrosofate; Fluorouracil; Cetuximab; Bevacizumab; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- irinotecan liposome (II), fluorouracil in combination with bevacizumab (Experimental): Experimental: irinotecan liposome (II), fluorouracil in combination with bevacizumab Induction therapy: irinotecan liposome (II), fluorouracil in combination with bevacizumab Maintenance therapy: bevacizumab with irinotecan liposome (II) or Capecitabine
  Interventions: Drug: irinotecan liposome (II); Drug: fluorouracil; Drug: bevacizumab; Drug: Capecitabine
- irinotecan liposome (II), fluorouracil in combination with cetuximab (Experimental): Experimental: irinotecan liposome (II), fluorouracil in combination with cetuximab Induction therapy: irinotecan liposome (II), fluorouracil in combination with bevacizumab Maintenance therapy: cetuximab with irinotecan liposome (II) or Capecitabine
  Interventions: Drug: irinotecan liposome (II); Drug: fluorouracil; Drug: cetuximab; Drug: Capecitabine

INTERVENTIONS:
Drug: irinotecan liposome (II) — irinotecan liposome (II) is a powerful chemotherapeutic agents, in the combination with fluorouracil，and bevacizumab or cetuximab
  Other Names: irinotecan liposome (II) injection
Drug: fluorouracil — fluorouracil is a powerful chemotherapeutic agents, in the combination with irinotecan liposome (II)，and bevacizumab or cetuximab
  Other Names: 5-fluorouracil
Drug: cetuximab — cetuximab is a powerful targeted agents, in the combination with irinotecan liposome (II)，and fluorouracil
  Other Names: cetuximab injection
  Arms: irinotecan liposome (II), fluorouracil in combination with cetuximab
Drug: bevacizumab — bevacizumab is a powerful targeted agents, in the combination with irinotecan liposome (II)，and fluorouracil
  Other Names: bevacizumab injection
  Arms: irinotecan liposome (II), fluorouracil in combination with bevacizumab
Drug: Capecitabine — Capecitabine is a powerful chemotherapeutic agent, in the combination with bevacizumab or cetuximab

SUMMARY:
Guidelines recommend FOLFIRI in combination with bevacizumab or cetuximab as a treatment option for advanced second-line colorectal cancer, and this study explores the efficacy and safety of a clinical study of liposomal irinotecan (II), fluorouracil, in combination with bevacizumab or cetuximab for the second-line treatment of patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
Guidelines recommend FOLFIRI in combination with bevacizumab or cetuximab as a treatment option for advanced second-line colorectal cancer. Liposomal irinotecan (II) compared with ordinary irinotecan can improve efficacy and safety. This study explores the efficacy and safety of a clinical study of liposomal irinotecan (II), fluorouracil, in combination with bevacizumab or cetuximab for the second-line treatment of patients with advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent to voluntarily enroll in this study.
2. Men or women aged 18-75 years.
3. Histologically or cytologically confirmed metastatic colorectal adenocarcinoma.
4. Patients who have failed one prior systemic therapy.
5. Eastern Cooperative Oncology Group Performance Status score of 0 or 1.
6. Life expectancy of at least 3 months.
7. Measurable lesions at baseline as assessed by the investigator by imaging (according to RECIST 1.1), measurable lesions should not have received local treatment such as radiotherapy (lesions located within the area of previous radiotherapy may also be selected as target lesions if progression is confirmed to have occurred).
8. Function of vital organs in accordance with the following requirements (no medication with any blood component, cell growth factor corrective therapy is allowed within 14 days prior to the first administration of study drug); Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Platelets ≥ 100 x 109/L; Haemoglobin ≥ 9 g/dL; Serum albumin ≥ 2.5 g/dL; Total bilirubin ≤ 1.5 × upper limit of normal; alanine aminotransferase, aspartate aminotransferase≤ 2.5 × upper limit of normal, and if liver metastases are present, alanine aminotransferase, aspartate aminotransferase ≤ 5 × upper limit of normal Serum creatinine ≤ 1.5 × upper limit of normal or creatinine clearance > 60 mL/min (Cockcroft-Gault); Activated partial thromboplastin time (APTT) and International Normalised Ratio (INR) ≤ 1.5 × upper limit of normal (screened for use of stable doses of anticoagulant therapy such as low molecular heparin or warfarin where the INR is within the expected therapeutic range of the anticoagulant).
9. Female subjects of childbearing potential must have a negative serum pregnancy test within 72 hours prior to initiation of trial drug administration and use effective contraception (e.g., intrauterine device, birth control pills, or condoms) during the trial period and for at least 3 months after the last dose of trial drug; for male subjects whose partner is a female of childbearing potential, effective contraception should be used during the trial period and for at least 3 months after the last dose of trial drug. For male subjects whose partners are women of childbearing potential

Exclusion Criteria:

1. Have received local radiotherapy within 4 weeks prior to the first dose of study drug and have not recovered to baseline levels of adverse events due to radiotherapy. Subjects who have had palliative radiotherapy to a peripheral site (e.g., bone metastases) prior to 4 weeks may be admitted to the study, provided they have recovered from any acute adverse events;
2. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects previously treated for brain metastases may enter the study provided they have stable brain metastases and have not been treated for brain metastases with steroids for at least 28 days prior to study entry. This exception does not include carcinomatous meningitis, as patients with carcinomatous meningitis are excluded regardless of clinical stability;
3. Major surgery, open biopsy, or severe trauma 28 days prior to first dose;
4. Have a previous history of hypersensitivity to fluorouracil or irinotecan;
5. Subjects with hypertension that is not well controlled with antihypertensive medication (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg)
6. Subject has uncontrolled cardiovascular clinical symptoms or disease, including but not limited to: (1) New York Heart Association Class II or higher heart failure (2) unstable angina (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmia that is not clinically interfered with or remains poorly controlled after clinical intervention.
7. Clinically significant bleeding symptoms or a definite bleeding tendency within 3 months prior to the first dose, e.g., gastrointestinal bleeding, bleeding gastric ulcer, or vasculitis;
8. Arterial/venous thrombotic events within 6 months prior to the first dose, such as cerebrovascular accidents (including temporary ischaemic attack, cerebral haemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, with superficial venous thrombosis being eligible for enrolment as determined by the investigator;
9. Have another malignancy that is progressing or requires aggressive treatment, except for non-melanoma skin cancer and cervical cancer in situ for which potential treatment has been administered;
10. Women who are pregnant or breastfeeding;
11. Subjects who, in the judgement of the investigator, have other factors that may cause them to be forced to terminate the study midway, such as other serious illnesses (including psychiatric illnesses) that require comorbid treatment, grossly abnormal laboratory test values, and family or social factors that may affect the subject's safety or the collection of trial data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | through study completion, an average of 1 year.
  Objective Response Rate

SECONDARY OUTCOMES:
Progression-free survival | median progression-Free-Survival approximately 4-7 months
  Progression-Free-Survival
Overall survival | median overall survival approximately 8-20 months
  Overall survival
Adverse Events | through study completion, assessed up to 50 months
  All adverse medical events occurring after the subject has received the experimental All adverse medical events occurring after the subject has received the experimental intervention
Qol | through study completion, assessed up to 50 months
  Assessment of patients' quality of life by means of quality of life score questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No